CLINICAL TRIAL: NCT04825548
Title: Post-thrombotic Syndrome After Deep Venous Thrombosis (DVT) in Patients Treated According to the NOPHO ALL2008 Protocol
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, M.D., PhD, Associate Professor, Aarhus University Hospital
Other Study IDs: PTS-NOPHOALL2008
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Acute Lymphoblastic Leukemia; Post Thrombotic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Examination of patients with previous DVT

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common malignant disease in childhood. Today more than 90% of children and 75% of adults (18-45 years) survive ALL. The enzyme Asparaginase (Asp) is an indispensable part of the multiagent treatment of ALL.

Treatment related severe acute toxicities are common. Especially in teenagers and adults, thromboembolism is one of the most common acute toxicities and may result in post thrombotic syndrome (PTS) or pulmonary hypertension. The knowledge about these late effects is limited, including for ALL patients.

ELIGIBILITY:
Inclusion Criteria:

* Treated on the ALL2008 protocol for ALL. Had a DVT on treatment.

Exclusion Criteria:

* Death

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients between 1.0-45 years of age and diagnosed with DVT and PE during treatment on the NOPHO ALL2008 protocol. In this period, 115 patients were diagnosed with DVT
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with post thrombotic syndrome | 01112020-01022023

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Vælg En Region, Stat Eller Provins., Denmark